CLINICAL TRIAL: NCT02745756
Title: A Combined Cell Therapy Approach to the Treatment of Neuroblastoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no enrollment
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17181
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Neuroblastoma; Neoplasms, Nerve Tissue
Keywords: Children; Cancer; High-risk neuroblastoma
MeSH Terms: conditions — Neuroblastoma; Neoplasms, Nerve Tissue; Neoplasms | interventions — Stem Cell Transplantation; keyhole-limpet hemocyanin; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined Cell Therapy (Experimental): Hematopoietic progenitor cell (HPC) transplant (HPCT) with autologous tumor cell lysate and keyhole limpet hemocyanin (KLH) pulsed dendritic cell (DC) vaccine.
  Interventions: Procedure: Autologous Hematopoietic Progenitor Cell Transplant; Biological: KLH and Tumor Lysate Pulsed DC Vaccine

INTERVENTIONS:
Procedure: Autologous Hematopoietic Progenitor Cell Transplant — Autologous Hematopoietic Progenitor Cell (HPC) Transplant (HPCT). Blood stem cells will be collected by apheresis during the induction phase as part of standard treatment. During apheresis, the participant's blood is collected into a machine that filters out the stem cells and the filtered blood is returned to their body. The stem cells will be separated by the type of protein within the cells. Only the stem cells with a protein called CD34 will be used for the stem cell transplant.
  Other Names: stem cell transplant
Biological: KLH and Tumor Lysate Pulsed DC Vaccine — Keyhole limpet hemocyanin (KLH) pulsed dendritic cell (DC) vaccine. Post-transplant vaccine days: +14, +28, +56 (± 10 days), +84 (± 10 days). Vaccines will be administered by intradermal injection of 0.5 mL at two nodal basins.
  Other Names: Dendritic Cell (DC) Vaccine

SUMMARY:
This study adds an experimental treatment with another type of cells, called dendritic cells. It is hoped that these cells may stimulate the immune system to react against neuroblastoma in much the same way that vaccines cause the immune system to react to certain viruses and bacteria. The physicians conducting this study have observed from previous research that neuroblastoma cells can be recognized by the immune system, and that they can be destroyed by immune cells.The main goal of this study is to see if giving participants this additional anti-Neuroblastoma vaccine reduces the risk of relapse following the Hematopoietic Stem Cell Transplant.

DETAILED DESCRIPTION:
All patients who are enrolled in this study will receive all treatment at All Children's Hospital which is located at 501 6th Ave South, St. Petersburg, FL 33701. This includes autologous cell donation by apheresis, high dose cytotoxic therapy conditioning for autologous HPC transplant, post-transplant follow-up care, and all administration of dendritic cell vaccines and blood draws for post therapy immunological monitoring.

All preparation of cellular products, including hematopoietic progenitor cell products for autologous transplantation, and dendritic cell vaccine products, will be carried out in the Cell Therapy Facility located within the Moffitt Cancer Center, which is located at 12902 Magnolia Drive, Tampa, FL 33612.

ELIGIBILITY:
Inclusion Criteria:

* Must have a histological diagnosis of neuroblastoma or ganglioneuroblastoma and be either newly diagnosed with high risk disease or have failed previous treatment: Patients who have failed previous treatment may have had no more than one earlier autologous HPC transplant.
* Participant is expected to undergo autologous HPC transplantation that is consistent with standard of care.
* Must have the presence of residual resectable disease for which surgery is clinically indicated, and will be performed at Johns Hopkins All Children's Hospital.

Exclusion Criteria:

* Not an eligible candidate for collection by apheresis or HPC transplant.
* History of autoimmune disorder or immune deficiency disorder.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-08-21 (Actual); Study Completion 2017-08-21 (Actual)

PRIMARY OUTCOMES:
Occurrence of Sufficient Tumor Cell Lysate and Dendritic Cells | Up to 1 year
  The feasibility of manufacturing both a hematopoietic progenitor cell graft and multiple tumor lysate pulsed dendritic cell vaccine treatments from the same starting apheresis product, culminating in delivery of the vaccines in the immediate period following myeloablative therapy and autologous hematopoietic progenitor cell transplant period (autoHPCT). For what fraction of eligible patients can sufficient tumor cell lysate and dendritic cells, necessary for the production of the dendritic cell vaccines, be obtained? From what fraction would it be possible to make additional vaccines?

SECONDARY OUTCOMES:
Occurrence of Dendritic Cell Related Adverse Events | Up to 1 year
  Toxicities resulting from the administration of dendritic cell vaccines in the immediate post hematopoietic cell graft period.

OTHER OUTCOMES:
Rate of Anti-tumor Effect | Up to 1 year
  Whether a discernable anti-tumor effect resulting from autoHPCT therapy combined with dendritic cell vaccine therapy can be detected, either through monitoring of the patient's immune system for evidence of tumor specific immunity, or by monitoring for measureable clinical responses.

CONTACTS AND LOCATIONS:
Overall Officials: Shari Pilon-Thomas, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Gregory Hale, M.D., Principal Investigator — Johns Hopkins All Children's Hospital